CLINICAL TRIAL: NCT03111381
Title: Toradol to Reduce Ureteroscopic Symptoms Trial
Acronym: TRUST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000020245
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-08

CONDITIONS: Urinary Lithiasis; Kidney Diseases; Kidney Stone; Pain, Postoperative
MeSH Terms: conditions — Urolithiasis; Kidney Diseases; Kidney Calculi; Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group in this study will receive a one-time dose of Ketorolac 30mg intravenously after undergoing general anesthesia. Because the participants will be under general anesthesia, they will not know if they received the medication. The surgeon will also be blinded to this. The anesthesiologist will not be blinded as he/she will deliver the agent and because the use of Toradol may alter their usage of other intra-operative agents and post-operative agents
  Interventions: Drug: Toradol
- Non-Intervention Group (No Intervention): In the no-treatment group, participants will not receive a dose of intra-operative Ketorolac.

INTERVENTIONS:
Drug: Toradol — IV toradol
  Arms: Intervention Group

SUMMARY:
Double blinded randomized controlled clinical trial to assess the impact of intraoperative Toradol on post-operative pain scores for patients undergoing ureteroscopy for urinary stone management.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-center, prospective randomized clinical trial evaluating the efficacy of intraoperative Ketorolac on post-operative pain in patients undergoing ureteroscopy at Yale-New Haven Hospital.

The study population will include anyone between the age of 18-80 who is undergoing elective ureteroscopy for management of stone disease without contraindication to ketorolac.

Patients who are being consented to undergo a ureteroscopy with the PI will be asked to participate in this study. There is currently no consensus on standard of care regarding intraoperative analgesia for ureteroscopy. There is wide variability in practice, some clinicians choose to administer intraoperative analgesia while others rely only on the sedation effects of general anesthesia. This study is being carried out to see if administration of Ketorolac during ureteroscopy provides a post-operative benefit in pain scores when compared to no treatment.

The intervention group in this study will receive a one-time dose of Ketorolac 30mg intravenously after undergoing general anesthesia. Because participants will be under general anesthesia, participants will not know if they received the medication. Following the procedure, the intervention group may continue to use Ketorolac as needed to manage pain. The only difference between the intervention group and the non-intervention group is the one time dose of intraoperative ketorolac.

The FDA approves Ketorolac as a nonsteroidal anti-inflammatory drug (NSAID), indicated for the short-term (up to 5 days in adults) management of moderately severe acute pain that requires analgesia at the opioid level.

Following assessment of eligibility and documentation of consent to participate in the study, participants will be randomized to receive intraoperative Ketorolac Tromethamine (Toradol®) or not. In the no-treatment group, participants will not receive a dose of intra-operative Ketorolac. Pain will be managed in the standard way with post-operative Ketorolac as needed. In the treatment group, participants will receive one dose of Ketorolac IV 30mg during the procedure. Randomization will occur by the attending anesthesiologist.

For this trial, the investigators, surgical team, and patients will be blinded to the administration of the agent, which is given as an IV Push of 30mg. For patients who are older than 65 years or weight less than 50kg, the dose will be adjusted to 15mg to minimize the risk of bleeding. The anesthesiologist will not be blinded as he/she will deliver the agent and because the use of ketorolac may alter their usage of other intra-operative agents and post-operative agents. The surgical team will be un-blinded post-operatively.

Following the procedure, participants will rate their pain using a visual pain assessment scale at 1 hour postoperatively and at the time of discharge from the recovery room. Once the patient is at home, the participant will fill out a validated survey that has questions related to pain. This will be filled out once a day for a total of 7 days following the procedure. In addition, the investigators will provide a medication utilization diary sheet for the participant to record daily use of prescribed narcotic and other as needed over the counter medications such as acetaminophen and ibuprofen.This will also be done daily for a total of 7 days. The participant will be surveyed at a one-week postoperative visit using the same assessment. All adverse drug reactions will be recorded from the time of administration to initial follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Ureteroscopy for kidney stone management between age 18-80.

Exclusion Criteria:

* Unable to provide consent
* Contraindications to Toradol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Medial Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Non-Intervention Group
Started | 46 | 48
Completed | 46 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Non-Intervention Group | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (147) | 33 (147) | 33 (146)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 23 | 26 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Once the patient is at home, they will fill out a validated visual analog pain scale to rate their pain. This will be filled out once a day for a total of 7 days following the procedure.
  This is total morphine equivalent use. The range is 0 to infinity. Higher scores are equated to worse pain. The units are "ME" or morphine equivalents.
Time Frame: up to 1 week
Measure: Mean (Standard Deviation); unit: milligram morphine equivalent
Arm/Group | Intervention Group | Non-Intervention Group
Number analyzed (Participants) | 46 | 48
milligram morphine equivalent | 22 (14) | 30 (18)

2. Secondary Outcome: Number of Participants With Complications
Time Frame: 6 weeks post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Non-Intervention Group
Number analyzed (Participants) | 46 | 48
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for 30 days from time of surgery
Arm/Group | Intervention Group | Non-Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT03111381/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT03111381/ICF_001.pdf